CLINICAL TRIAL: NCT05670470
Title: A Prospective, Randomized, Investigator-blinded, Parallel, Multi-center, Phase 3 Trial in Bowel Preparation for Colonoscopy
Brief Title: A Prospective, Randomized, Investigator-blinded, Parallel, Multi-center, Phase 3 Trial
Acronym: PROPELLER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taejoon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTP0303
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-01

CONDITIONS: Bowel Preparation
Keywords: Bowel Preparation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTP0303 (Experimental)
  Interventions: Drug: CTP0303
- Orafang Tab (Active Comparator)
  Interventions: Drug: Orafang Tab

INTERVENTIONS:
Drug: CTP0303 — Subjects who are randomized into group CTP0303 will receive bowel preparation from evening to next morning.
  Arms: CTP0303
Drug: Orafang Tab — Subjects who are randomized into group Orafang Tab will receive bowel preparation from evening to next morning.
  Arms: Orafang Tab

SUMMARY:
This is a prospective randomized study compared with active control arm.

DETAILED DESCRIPTION:
This is a prospective randomized study compared with active control arm. The investigators compare the colon cleansing in patients undergoing colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients and inpatients aged: ≥19
* A prospective colonoscopy person
* Written informed consent to participate in the trial

Exclusion Criteria:

* Patients with past history of severe constipation (requiring repeated use of laxatives/enema or physical intervention before resolution), known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or megacolon.
* Patients with ongoing severe acute Inflammatory Bowel Disease
* Patients who have had previous significant gastrointestinal surgeries, including colonic resection, subtotal colectomy, abdominoperineal resection, defunctioning colostomy, Hartmann's procedure and defunctioning ileostomy or other similar surgeries involving structure and function of the small or large colon.
* Pregnant women or pregnant women or pregnant women
* Patients who have not been confirmed to have COVID-19 for a month
* Severe heart disease (cardiac failure (NYHA class 3 and 4))
* Acute coronary artery disease within 24 weeks before screening (an unstable angina pectoris, acute myocardial infarction), clinically significant arrhythmia, hypertrophic obstruction Cardiomyopathy, valvular disease, aortic and peripheral vascular diseases
* Patients with severe chronic renal impairment (glomerular filtration rate less than 30ml/min/1.73m2)
* People who have hypersensitivity or allergies to clinical trial drug components

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Number of Patients With Successful Bowel Cleansing (Overall Colon) | 1 day of scheduled colonoscopy
  The overall quality of bowel cleansing was assessed by a blinded central reader (an experienced and trained colonoscopist) using the segmental scores of the Harefield Cleansing Scale (HCS). A final HCS grading of A, B, C or D was derived. Grades A and B are classified as successful (i.e. all mucosa could be visualized) and C and D are classified as unsuccessful.

SECONDARY OUTCOMES:
Number of Patients With 'Excellent Plus Good' (Highly Effective) Bowel Cleansing (Colon Ascendens) | 1 day of scheduled colonoscopy
  The overall quality of bowel cleansing was assessed by a blinded central reader (an experienced and trained colonoscopist) using the segmental scores of the Harefield Cleansing Scale (HCS). Highly effective cleansing in the colon ascendens corresponded to scores 3 (Good) or 4 (Excellent) of the HCS.
Adenoma/Polyp Detection Rate (Overall Colon) | 1 day of scheduled colonoscopy
  Through colonoscopy, a blinded central reader checks whether polyp or adenoma is found, and if more than one polyp or adenoma is found in a patient, it is defined as "detection." The polyp detection rate (PDR) and adenoma detection rate (ADR) of the entire colon and ascending colon are defined as follows.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Myung Cha, MD, PhD, Principal Investigator — Kyung Hee University Hospital at Gangdong
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, Gangdong, South Korea

REFERENCES:
- [Derived] Jeon SR, Park SK, Yang DH, Cha JM. Comparison of a novel mini-oral sulfate tablet and the conventional oral sulfate tablet in bowel preparation for colonoscopy: a prospective, randomized, investigator-blinded, multicenter, non-inferior, phase 3 trial. J Gastroenterol. 2023 Nov;58(11):1114-1123. doi: 10.1007/s00535-023-02023-5. Epub 2023 Aug 5. PMID 37542674